CLINICAL TRIAL: NCT06907407
Title: Effect Of Different Diaphragmatic Myofascial Release Approaches On Low Back Pain And Quality Of Life Among Young Females With Irritable Bowel Syndrome
Acronym: IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Noha Hamdy Abd El-Khaleq Teama, principle investigator : noha hamdy abd elkhaleq, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003707
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Irritable Bowel Syndrome
Keywords: Diaphragmatic Myofascial Release; Low Back Pain; Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome; Low Back Pain

STUDY DESIGN:
Intervention Model Description: diaphragmatic myofascial release and visceral mobilization
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelope
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diaphragmatic Myofascial Release (Experimental): thirty female will receive diaphragmatic breathing exercise, different diaphragmatic myofascial release approaches, visceral mobilization techniques, irritable bowel syndrome medication under supervision of a physician for 50 minutes twice a week for 4 weeks
  Interventions: Other: Diaphragmatic Myofascial Release; Other: irritable bowel syndrome medication
- visceral mobilization techniques (Experimental): thirty female will receive visceral mobilization techniques and irritable bowel syndrome medication under supervision of a physician for 50 minutes twice a week for 4 weeks
  Interventions: Other: visceral mobilization techniques; Other: irritable bowel syndrome medication
- irritable bowel syndrome medication (Active Comparator): thirty female will receive irritable bowel syndrome medication under supervision of a physician for 50 minutes twice a week for 4 weeks
  Interventions: Other: irritable bowel syndrome medication

INTERVENTIONS:
Other: Diaphragmatic Myofascial Release — six technique will be applied; 1-Diaphragmatic transverse plane, 2-Anteroposterior equilibrium technique, 3-Supra and infrahyoid fascial induction, 4-Psoas fascial induction,5-Diaphragm stretching technique and 6-Phrenic centre inhibition. diaphragmatic breathing, Mobilization of the ascending colon, descending colon, sigmoid colon, and sphincters (cardiac, pyloric, Oddi, duodenojejunal and ileocecal) with the patient in the supine position, knees flexed, feet supported and abdomen exposed. Contact was made with the region to be treated, leading it in the direction of immobility, with pressure maintained for one minute on each region with intensity based on the sensitivity to tension observed on the feedback of the individual plus medication
  Arms: Diaphragmatic Myofascial Release
Other: visceral mobilization techniques — Mobilization of the ascending colon, descending colon, sigmoid colon, and sphincters (cardiac, pyloric, Oddi, duodenojejunal and ileocecal) with the patient in the supine position, knees flexed, feet supported and abdomen exposed. Contact was made with the region to be treated, leading it in the direction of immobility, with pressure maintained for one minute on each region with intensity based on the sensitivity to tension observed on the feedback of the individual plus medication
  Arms: visceral mobilization techniques
Other: irritable bowel syndrome medication — the patients will receive irritable bowel syndrome medication

SUMMARY:
this study will be conducted to investigate the effect of different diaphragmatic myofascial release approaches on low back pain and quality of life among young females with irritable bowel syndrome

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is a functional gastrointestinal disorder linked to disruptions in autonomic nervous system regulation, gut inflammation, alterations in stool frequency, and visceral hypersensitivity. Irritable bowel syndrome (IBS) is a chronic condition affects 7 to 21% of the general population.The symptoms usually include abdominal cramping, discomfort or pain, bloating, loose or frequent stools and constipation.The diaphragm has a fundamental role in defining posture, its maintenance, and body position changes; dysfunction of the diaphragm is one of the recognized be causes of low back and sacroiliac joint pain. People with low back pain often experience early fatigue of the diaphragm muscle, altered and reduced excursion during respiration, and inadequate proprioceptive activation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with irritable bowel syndrome
* Young female subjects
* All patients will have low back pain.
* All subjects will be clinically and medically stable when attending the study

Exclusion Criteria:

* Lack of attention and cooperation
* History of cancer and any systemic disease
* Pregnancy
* History of any structural gastrointestinal pathology or surgery
* History of repeated inflammatory gastrointestinal pathology
* Diabetes mellitus and lactose intolerance.
* Abuse of laxative
* Depression
* Celiac disease
* Endocrine disorders as hypothyroidism and hyperthyroidism.
* Gastrinoma
* Recent/unhealed rib fracture
* History of any lumbar spine serious pathology ( tumor, infection fracture, osteoporosis , long term use of steroid, rheumatoid arthritis and surgery )

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Lumbar spine mobility | up to four weeks
  shober's test will be used to assess sine mobility. • Patient is standing, examiner marks on the midpoint between the posterior superior iliac spines by drawing a horizontal line across the patient's back. a second line is marked 10 cm above the first line. Patient is then instructed to flex forward as if attempting to touch his/her toes, examiner remeasures distance between two lines with patient fully flexed. The difference between the measurements in erect and flexion positions indicates the outcome of the lumbar flexion Elongation of 5 cm or more between the two marks during forward flexion is considered to be normal lumbar spine movement
low back disability | up to four weeks
  The Oswestry Disability Index will be used.It is self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for one self, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel, Each section is scored on a 0-5 scale, 5 representing the greatest disability. The index is calculated by dividing the summed score by the total possible score, which is then multiplied by 100 and expressed as a percentage. Thus, for every question not answered, the denominator is reduced by 5. If a patient marks more than one statement in a question, the highest scoring statement is recorded as a true indication of disability. Then the score classified into mild 5 -14, moderate 15-24, sever 25-34, disabled 35 -50 The questionnaire takes 3.5-5 min to complete and approximately 1 min to score

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Giza, Egypt